CLINICAL TRIAL: NCT06196658
Title: Early Phase I Study of Autologous T Cells Engineered to Express Anti-EX02 Chimeric Antigen Receptor (EX02 CAR-T) for Unresectable Pancreatic/Bile Duct Cancer
Brief Title: Early Phase I Study of Autologous T Cells (EX02 CAR-T) for Unresectable Pancreatic/Bile Duct Cancer
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhang Xiaofeng,MD (Other)
Collaborators: Zeno Therapeutics Pte. Ltd (Unknown)
Responsible Party: Sponsor-Investigator, Zhang Xiaofeng,MD, chief physician, First People's Hospital of Hangzhou
Organization: First People's Hospital of Hangzhou (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20231226
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Pancreatic Cancer; Advanced Biliary Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-EX02 CAR T cells (Experimental)
  Interventions: Drug: anti-EX02 CAR T cells

INTERVENTIONS:
Drug: anti-EX02 CAR T cells — Conditioning chemotherapy:
  • Lymphodepletion regimen consisting of fludarabine 25 mg/m2/day and cyclophosphamide 250 mg/m2/day for 3 consecutive days, administered 48 hours before first administration of first time of intravenous or intraperitoneal infusion
  Investigational Product:
  • Regional administration: Acetaminophen 500mg orally and diphenhydramine 20mg intramuscularly (or other non-steroidal anti-inflammatory drugs and antihistamines) were given in advance on the day of administration (day 0). Intraperitoneal infusion or intra-tumoral injection of anti-EX02 CAR T cells, with dosage and method determined by the investigator
  • Intravenous administration: Single infusion of CAR-transduced autologous T cells administered intravenously at a target dose of 2 x 106 anti-EX02 CAR T cells/kg, 30 minutes after premedication with oral acetaminophen 500mg and intramuscular diphenhydramine 20mg

SUMMARY:
This is a early Phase 1 open-label study to explore the safety and possible efficacy of EX02 CAR T cell therapy in the treatment of patients with unresectable and/or metastatic pancreatic/bile duct cancer.

Each participant will undergo leukapheresis after enrolment, receive treatment of the conditioning chemotherapy of cyclophosphamide and fludarabine, and an intra-tumoral injection or intraperitoneal infusion of Ex02 CAR T cells, probably followed by an intravenous infusion of EX02 CAR T cells.

Each participant will proceed through the following study procedures:

* Screening
* Enrollment/Leukapheresis
* Conditioning chemotherapy
* CAR T treatment
* Post-treatment assessment
* Long-term follow-up

ELIGIBILITY:
Inclusion Criteria:

* 1) Must have a confirmed diagnosis of unresectable or metastatic pancreatic cancer or bile duct cancer 2) Ineligible for, refractory to or relapsed after first or second line of chemotherapy 3) Presence of at least one measurable target lesion according to RECIST v1.1 4) EX02 positive tumor cell membrane (as shown in IHC staining of tumor specimen or in flow cytometry of ascites cells) 5) Male or female, ≥18 years 6) ECOG performance status 0 to 1 7) Expected life expectancy >3 months 8) Negative pregnancy test at screening and prior to initiating lymphodepletion chemotherapy or study drug administration, and willingness to practice birth control for woman with childbearing potential 9) Adequate hematology function indicated by followings (without blood transfusion or administration with growth factors in last four weeks):

  1. Neutrophil count ≥ 1.5×10^9/L
  2. Hemoglobin ≥ 90g/L
  3. Platelet count ≥ 100×10^9/L
  4. Lymphocyte count ≥ 0.5×10^9/L 10) Adequate liver, kidney, heart and lung functions at least indicated by:

  <!-- -->

  1. Creatinine clearance ≥ 60ml/min
  2. ALT and AST ≤ 2.5 ULN (≤ 5 ULN when liver is involved)
  3. LVEF ≥ 50%; absence of pericardial fluid; no significant abnormality in ECG exam
  4. No or only small amount of pleural fluid or ascites; blood oxygen saturation ≥ 95% 11) Voluntary participation in the trial and signing informed consent form

Exclusion Criteria:

* 28 participants fulfilling the following criteria will be enrolled.

Inclusion criteria:

1. Must have a confirmed diagnosis of unresectable or metastatic pancreatic cancer or bile duct cancer
2. Ineligible for, refractory to or relapsed after first or second line of chemotherapy
3. Presence of at least one measurable target lesion according to RECIST v1.1
4. EX02 positive tumor cell membrane (as shown in IHC staining of tumor specimen or in flow cytometry of ascites cells)
5. Male or female, ≥18 years
6. ECOG performance status 0 to 1
7. Expected life expectancy >3 months
8. Negative pregnancy test at screening and prior to initiating lymphodepletion chemotherapy or study drug administration, and willingness to practice birth control for woman with childbearing potential
9. Adequate hematology function indicated by followings (without blood transfusion or administration with growth factors in last four weeks):

   1. Neutrophil count ≥ 1.5×10^9/L
   2. Hemoglobin ≥ 90g/L
   3. Platelet count ≥ 100×10^9/L
   4. Lymphocyte count ≥ 0.5×10^9/L
10. Adequate liver, kidney, heart and lung functions at least indicated by:

    1. Creatinine clearance ≥ 60ml/min
    2. ALT and AST ≤ 2.5 ULN (≤ 5 ULN when liver is involved)
    3. LVEF ≥ 50%; absence of pericardial fluid; no significant abnormality in ECG exam
    4. No or only small amount of pleural fluid or ascites; blood oxygen saturation ≥ 95%
11. Voluntary participation in the trial and signing informed consent form

Exclusion criteria:

1. Active viral infection including but not limiting hepatitis A, hepatitis B, hepatitis C or HIV
2. History of acquired immunodeficiency syndrome (AIDS)
3. Is pregnant or lactating
4. Unwilling to practice birth control
5. Planned intraperitoneal chemotherapy (such as HIPEC) within 28 days
6. Received systemic immune inhibitors or corticosteroids (prednisone 15mg/day or above equivalent dose) within 2 weeks of the time of initiating conditioning chemotherapy
7. Current involvement of:

   1. Active infection which requires treatment with systemic administration
   2. Active coagulation disorders or receiving anti-coagulant treatment (except for aspirin)
   3. Active hemolytic anemia
   4. Significant arrhythmia, or history of myocardial infarction, ventricular tachycardia, or ventricular fibrillation
   5. Active obstructive or constrictive lung disease
   6. Active autoimmune disease such as rheumatoid arthritis or immunodeficiency disease
   7. Active CNS metastases or cerebrospinal malignancy
   8. Uncontrolled diseases including disorders of cardiovascular, respiratory, renal, gastrointestinal, urogenital or immune systems
8. Active second malignancy in addition to the studied one, excluding low-risk neoplasms such as non-metastatic basal cell or squamous cell skin carcinoma
9. History of hypersensitivity to any drugs planning to be used in this study
10. History of treatment with any genetically modified T cell therapy (including CAR T cells and TCR T cells)
11. Any conditions that investigator consider as ineligibility of participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of treatment-related adverse events (TEAEs) | 4 weeks after the first CAR-T cell infusion
  Grade and type of toxicity per dose level; fraction of patients who experience toxicity (including allergic reactions to T cell infusions) of ≥ Grade 3 according to CTCAEv5.0, cytokine release syndrome (CRS) of ≥ Grade 3 according to ASTCT consensus and Immune Effector Cell-Associated Neurotoxicity Syndrome (ICANS).
Objective Response Rate | 24 weeks
  Objective Response Rate (ORR) is the proportion of participants with an objective response (either a complete response [CR] or partial response [PR]) in participants who received at least 1 dose of EX02CART and at least the 6-week tumor evaluation as determined by the investigator according to RECIST v1.1.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 24 weeks
  PFS is the time between the date of first dose and the date of first documented disease progression as determined by the investigator using RECIST v1.1 or death due to any cause, whichever occurs first.
Duration of Response (DOR) | 24 weeks
  DOR is the time from onset of response to progression or death due to any reason, whichever occurs first.
Overall survival (OS) | 24 weeks
  OS is the time between the date of first dose and the date of death due to any reason.
Disease control rate (DOC) | 24 weeks
  DOC is the proportion of participants with a stable disease (SD) or an objective response (CR or PR) in participants who received at least 1 dose of EX02CART and at least the 6-week tumor evaluation as determined by the investigator according to RECIST v1.1.
5) Volume of ascites measured by ultrasonography and/or frequency and volume of ascites aspiration | 24 weeks

IPD SHARING:
Plan to Share IPD: No